CLINICAL TRIAL: NCT01954693
Title: TRON: A Randomised, Double Blind, Placebo-controlled Study of RAD001 (Everolimus) in the Treatment of Neurocognitive Problems in Tuberous Sclerosis
Brief Title: A Study of Everolimus in the Treatment of Neurocognitive Problems in Tuberous Sclerosis
Acronym: TRON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiff University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Julian Sampson, Professor, Cardiff University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPON803-10; 2011-004854-25 (EudraCT Number)
Record Dates: First submitted 2013-09-05; First posted 2013-10-07 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Tuberous Sclerosis
Keywords: Tuberous Sclerosis; Everolimus; Neurocognitive functioning
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (RAD001) (Experimental): 2x2.5mg daily
  Interventions: Drug: Everolimus (RAD001)
- Placebo (Placebo Comparator): 2x2.5mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 5mg daily administered for 6 months as two oral 2.5 mg tablets once daily.
  Arms: Placebo
Drug: Everolimus (RAD001) — 5mg daily administered for 6 months as two oral 2.5 mg tablets once daily
  Arms: Everolimus (RAD001)

SUMMARY:
This is a single centre, two-arm, individually randomised, Phase II, double- blind, placebo-controlled trial of RAD001 (Everolimus) versus placebo in the treatment of neurocognitive problems in patients with tuberous sclerosis (TSC). The IMP is a licensed medicine in this patient group but for a different target of effect. The current trial is a proof of principle study for memory and executive function outcomes.

Following an eligibility visit, patients will be scheduled for baseline visit and randomization. They will then be followed up for 6 months undergoing both safety and neurocognitive assessments whilst taking either the placebo or study drug.

48 patients aged 16 to 60 years with tuberous sclerosis (TSC) who have IQ > 60 and a significant deficit in one or more primary outcome measures will be randomly allocated in a ratio of 2:1 to either RAD001 (Everolimus) or Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Definite TSC by current clinical criteria (28);
2. Male or female aged 16 to 60 yrs;
3. IQ over 60 by Wechsler Abbreviated Scales of Intelligence (WASI) and able to participate in direct neuropsychological tests;
4. A score falling on, or below, the 5th percentile (approximately equivalent to -1.5 SD) in one or more of the primary outcome measures:
5. Calculated GFR > 60ml/min/1.73m2 except in case of renal impairment associated with TSC complicating kidneys, where a calculated GFR should be ≥30ml/min/1.73m2;
6. INR 1.5 or less (anticoagulation permitted if target INR on stable dose of warfarin or LMW heparin for > 2 weeks at time of randomisation) ;
7. Adequate liver function as shown by: serum bilirubin less than or equal to 1.5 x ULN, ALT and AST less than or equal to 2.5 x ULN;
8. If sexually active - negative pregnancy test in females at the time of informed consent, contraception for males and pre-menopausal females on study);
9. Seizure free or stable seizures as defined by no change in type of AEDs in 6 months prior to full recruitment and randomization at baseline. Doses of drugs may have been changed in the 6 months prior to recruitment;
10. Hepatitis B surface antigen negative, Hepatitis C antibody negative.
11. All patients must be able to communicate well with the investigator, to understand and comply with the requirements of the study, understand and sign the written informed consent;
12. Female patients of childbearing potential must be prepared to use two acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.), from the time of screening.

Exclusion Criteria:

1. Prior treatment with an mTOR inhibitor;
2. Investigational agent <30 days prior to randomisation;
3. Surgery in last 2 months;
4. Previous brain neurosurgery;
5. Significant haematological abnormality i.e. haemoglobin < 8g/dL, platelets <80,000/mm3, absolute neutrophil count < 1000/mm3);
6. Urine protein/creatinine >0.02g/mmol except in case of renal impairment associated with TSC complication of kidneys, where urine protein/creatinine ratio should be >0.1g/mmol for exclusion;
7. Serum creatinine > 1.5 x ULN except in case of renal impairment associated with TSC complication of kidneys, where serum creatinine should be >300µmol/L for exclusion;
8. Uncontrolled hyperlipidaemia (fasting cholesterol > 300mg/dL or >7.75 mmol/L and fasting triglycerides >2.5 x ULN, or diabetes with fasting serum glucose > 1.5 x ULN;
9. History of myocardial infarction, angina or stroke related to atherosclerosis, or any other significant cardiac disease, HIV seropositivity, organ transplant, malignancy other than squamous or basal cell skin cancer;
10. lymphangioleiomyomatosis with FEV1 <70% of predicted, or any other restrictive pulmonary disease;
11. Bleeding diathesis or on oral anti-vitamin K medication other than low dose warfarin;
12. Pregnancy/lactation;
13. Live vaccine required during trial;
14. Use of strong inhibitor of CYP3AE;
15. Use of strong inducer of CYP3AE except for anti epileptic drugs;
16. Intercurrent infection at time of randomisation;
17. Inability to complete study materials (outcome measures) in English;
18. History of significant trauma-related cognitive deficit;
19. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of Everolimus (e.g. pancreatic insufficiency);
20. Known sensitivity to Everolimus or other Rapamycin analogues or to its excipients;
21. Inability to attend scheduled visits.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-06; Primary Completion 2018-08-06 (Estimated); Study Completion 2018-08-06 (Estimated)

PRIMARY OUTCOMES:
List Learning test (from the BIRT Memory and Information Processing Battery) | 6 months
Complex Figure test (from the BIRT Memory and Information Processing Battery) | 6 months
CANTAB - Stockings of Cambridge (SOC) | 6 months
CANTAB - Spatial Working Memory (SWM) | 6 months
Telephone search dual task (from the Test of Everyday Attention) | 6 months

SECONDARY OUTCOMES:
CANTAB - Rapid Visual Information Processing Battery (RVIP) | 6 months
CANTAB - Spatial Span (SSP) | 6 months
CANTAB - Attentional Set-shifting (IDED) | 6 month
Verbal Fluency /Controlled Oral Word Association Test (COWAT) | 6 months
Cancellation task | 6 months
Symptom Checklist 90R (SCL-90R) | 6 months
Quality of Life in Epilepsy (QOLIE) | 6 months
Liverpool Seizure Severity Scale (LSSS) | 6 months
Vineland Adaptive Behavior Scales-II (VABS-II) (survey form) | 6 months
Social Responsiveness Scale - Adult version (SRS-A) | 6 months
Social communication questionnaire (SCQ) | 6 months
National Adult Reading Test (NART) | 6 months

OTHER OUTCOMES:
Wechsler Abbreviated Scale of Intelligence (WASI) (4 subtests) | Eligibility visit
  Eligibility visit screening measure
Edinburgh Handedness Test | Eligibility visit
  Eligibility visit screening measures

CONTACTS AND LOCATIONS:
Overall Officials: Julian Sampson, Prof, Principal Investigator — Cardiff University
Locations (1):
- Cardiff University, Cardiff, United Kingdom